CLINICAL TRIAL: NCT01757340
Title: Calorie Restriction With Leucine Supplementation in Postmenopausal Women
Brief Title: Calorie Restriction With Leucine Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Ajinomoto Co., Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRL-201102153
Record Dates: First submitted 2012-12-14; First posted 2012-12-28 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Obesity; Menopause; Osteoporosis; Sarcopenia
MeSH Terms: conditions — Obesity; Osteoporosis; Sarcopenia | interventions — Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Weight maintenance (No Intervention): Weight maintenance with normal protein and leucine intake
- Weight loss with normal protein intake (Active Comparator)
  Interventions: Behavioral: Weight loss with normal protein and leucine intake
- Weight loss with leucine supplementation (Experimental)
  Interventions: Behavioral: Weight loss with protein/leucine supplementation

INTERVENTIONS:
Behavioral: Weight loss with normal protein and leucine intake — Goal of 8 to 10% weight loss while consuming the recommended daily allowance of protein (i.e, 0.8 grams of protein per kg body weight per day).
  Arms: Weight loss with normal protein intake
Behavioral: Weight loss with protein/leucine supplementation — Goal of 8 to 10% weight loss while consuming 150% of the recommended daily allowance of protein (i.e., 1.2 grams of protein per kg body weight per day) with the additional protein given in the form of whey protein, which has a high leucine content.
  Arms: Weight loss with leucine supplementation

SUMMARY:
The purpose of this study is to determine whether consuming additional leucine during calorie restriction induced weight loss has beneficial or harmful effects on multi-organ (liver, muscle, adipose tissue) insulin sensitivity, colonocyte proliferation rates, the gut microbiome, muscle mass and function, and bone mineral density in obese, postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Obese with body mass index (BMI) between 30 and 40 kg/m2
* Postmenopausal
* Sedentary (i.e., less than 1.5 hours of exercise per week)

Exclusion Criteria:

* Individuals with diabetes and/or uncontrolled hypertension
* Individuals with hepatitis B and/or C
* Individuals who smoke
* Individuals with an allergy to whey protein

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change in muscle mass | Baseline and at 10% weight loss in calorie restriction groups and ~6 to 7 months in the weight maintenance group
  We will measure total appendicular skeletal muscle mass by using dual-energy X-ray absorptiometry (DXA) and thigh muscle volume by magnetic resonance imaging (MRI)
Change in muscle strength | Baseline and at 10% weight loss in calorie restriction groups and ~6 to 7 months in the weight maintenance group
  We will evaluate muscle strength by administering maximum one repetition strength and isokinetic strength tests.
Change in bone mineral density and bone mineral content | Baseline and at 10% weight loss in calorie restriction groups and ~6 to 7 months in the weight maintenance group
  We will evaluate total bone mass and total body and regional bone mineral density by using dual X-ray energy absorptiometry (DXA).

SECONDARY OUTCOMES:
Change in skeletal muscle insulin sensitivity | Baseline and at 10% weight loss in calorie restriction groups and ~6 to 7 months in the weight maintenance group
  We will evaluate insulin sensitivity using the hyperinsulinemic-euglycemic clamp procedure in conjunction with stable isotope labeled tracer infusions
Change in bacterial populations found in the stool | Baseline and at 10% weight loss in calorie restriction groups and ~6 to 7 months in the weight maintenance group
Change in cell proliferation (growth) rates in the colon | Baseline and at 10% weight loss in calorie restriction groups and ~6 to 7 months in the weight maintenance group
  We will examine colon cell proliferation rates using stable isotope labelled tracer methods in conjunction with sigmoid colon biopsy samples
Determine the acute effect of leucine ingestion on skeletal muscle insulin sensitivity | Prior to starting the weight loss or maintenance intervention
  We will evaluate insulin sensitivity using the hyperinsulinemic-euglycemic clamp procedure in conjunction with stable isotope labeled tracer infusions
Determine the acute effect of leucine ingestion on muscle protein metabolism | Prior to starting the weight loss or maintenance intervention
  We will assess rates of muscle protein synthesis, breakdown and net protein balance using stable isotope labeled tracer methods during postabsorptive conditions and during insulin infusion with or without leucine ingestion.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Result] Smith GI, Yoshino J, Stromsdorfer KL, Klein SJ, Magkos F, Reeds DN, Klein S, Mittendorfer B. Protein Ingestion Induces Muscle Insulin Resistance Independent of Leucine-Mediated mTOR Activation. Diabetes. 2015 May;64(5):1555-63. doi: 10.2337/db14-1279. Epub 2014 Dec 4. PMID 25475435
- [Derived] Harris LLS, Smith GI, Patterson BW, Ramaswamy RS, Okunade AL, Kelly SC, Porter LC, Klein S, Yoshino J, Mittendorfer B. Alterations in 3-Hydroxyisobutyrate and FGF21 Metabolism Are Associated With Protein Ingestion-Induced Insulin Resistance. Diabetes. 2017 Jul;66(7):1871-1878. doi: 10.2337/db16-1475. Epub 2017 May 4. PMID 28473464